CLINICAL TRIAL: NCT04499586
Title: A Phase II Trial of Radiotherapy Combined With Raltitrexed and Irinotecan(CPT-11) in Patients With Metastatic or Locally Recurrent Colorectal Cancer
Brief Title: A Study of Radiotherapy Combined With Raltitrexed and Irinotecan in Metastatic or Locally Recurrent Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhu Ji, professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-R006
Record Dates: First submitted 2020-07-31; First posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Recurrent Colorectal Cancer
Keywords: Recurrent Colorectal Cancer; Irinotecan; Raltitrexed; Chemoradiotherapy
MeSH Terms: conditions — Colorectal Neoplasms | interventions — raltitrexed; Irinotecan

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Radiotherapy Combined With Raltitrexed and Irinotecan (Experimental): Each cycle lasts 3 weeks. Administration of Raltitrexed and Irinotecan weekly followed by a 2 week 'rest' period with no drug given. Raltitrexed is given by IV infusion at a dose of 3mg/m2. Irinotecan is given by IV infusion at a dose of 80mg/m2 (UGT1A1*28 6/6) or 65mg/m2 (UGT1A1*28 6/7).Radiation: 45-55Gy/25-30Fx
  Interventions: Combination Product: Radiotherapy Combined With Raltitrexed and Irinotecan

INTERVENTIONS:
Combination Product: Radiotherapy Combined With Raltitrexed and Irinotecan — Each cycle lasts 3 weeks. Raltitrexed: 3mg/m2 per week. Irinotecan : 80mg/m2 (UGT1A1*28 6/6) or 65mg/m2 (UGT1A1*28 6/7) per week. Radiation: 45-55Gy/25-30Fx

SUMMARY:
The study evaluates the effectiveness of radiotherapy combined with raltitrexed and irinotecan in treating patients who have metastatic or locally recurrent colorectal cancer that has not responded to fluorouracil. The patients will receive radiotherapy combined with raltitrexed and irinotecan, and then the surgeons will evaluate whether they should receive a surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven metastatic, advanced, or locally recurrent fluorouracil (5-FU) and oxaliplatin refractory adenocarcinoma of the colon or rectum; Progression of disease within 6 months of receiving adjuvant 5-FU and oxaliplatin chemotherapy OR Progression of disease during or following completion of 5-FU and oxaliplatin chemotherapy for metastatic disease
* Evaluable lesions with indications of radiotherapy
* No other metastatic lesions in the radiation field
* Karnofsky Performance Status>=70
* UGT1A1*28 6/6 or 6/7
* Subject blood routine and biochemical indicators meet the following criteria: hemoglobin ≥ 90g / L; absolute neutrophil count (ANC) ≥ 1.5 × 109 / L; Alanine transaminase (ALT), aspartate aminotransferase (AST) ≤ 2.5 times the upper limit of normal; alkaline phosphatase (ALP) ≤2.5 times the normal upper limit; serum total bilirubin <1.5 times the normal upper limit; serum creatinine <1 times the normal upper limit; serum albumin ≥ 30g / L
* Able to follow the protocol during the study period
* Sign the inform consent

Exclusion Criteria:

* Pregnant or breastfeeding women
* If there is an uncontrolled history of epilepsy, central nervous system disease or mental disorder, the investigator may determine that the clinical severity may hinder the signing of informed consent or affect the patient's oral medication compliance.
* Clinically severe (ie, active) heart disease, such as symptomatic coronary heart disease, New York Heart Association (NYHA) class II or more severe congestive heart failure or severe arrhythmia requiring medication intervention (see appendix 12), or a history of myocardial infarction in the last 12 months
* Organ transplantation requires immunosuppressive therapy
* Severe uncontrolled recurrent infections, or other serious uncontrolled concomitant diseases
* Anyone who is allergic to any research medication

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR(Objective Response Rate) includes CR(Complete Rate) and PR(Partial Rate) | 20 weeks

SECONDARY OUTCOMES:
DCR(Disease Control Rate) | 20 weeks
PFS(Progression Free Survival) | 24 months
the morbidity of hematological adverse events and diarrhea as assessed by CTCAE v4.0 | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Zhang, MD, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China